CLINICAL TRIAL: NCT00215540
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Assess the Safety and Efficacy of SURFAXIN® (Lucinactant), in Very Low Birth Weight (VLBW) Infants at Risk for Developing Bronchopulmonary Dysplasia
Brief Title: SURFAXIN® Treatment for Prevention of Bronchopulmonary Dysplasia (BPD) in Very Low Birth Weight (VLBW) Infants.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Concerns related to availability of drug product
Sponsor: Windtree Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KL4-BPD-01
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Results first posted 2012-06-13 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-05

CONDITIONS: Respiratory Distress Syndrome, Newborn; Premature Birth; Bronchopulmonary Dysplasia
Keywords: Double-blind; Low Birth Weight; Surfactant; Placebo-Controlled; Premature Birth
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth; Bronchopulmonary Dysplasia | interventions — lucinactant; Surface-Active Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SURFAXIN High Dose (Experimental): SURFAXIN (lucinactant) at 175 mg/kg
  Interventions: Drug: Lucinactant 175 mg/kg
- SURFAXIN Low Dose (Experimental): SURFAXIN (lucinactant) at 90 mg/kg
  Interventions: Drug: Lucinactant 90 mg/kg
- Placebo (Placebo Comparator): Sham air using 3.0 mL/kg volume of air
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lucinactant 175 mg/kg — Administered via slow intra-tracheal instillation at a dose of 175 mg/kg (5.8 mL/kg of a 30-mg/mL suspension). Initial treatment given no later than 1 hour after randomization. Additional treatments were administered every 48 hours up to a maximum of 5 doses (up to day of life (DOL) 18).
  Other Names: SURFAXIN; Lucinactant; Surfactant
  Arms: SURFAXIN High Dose
Drug: Lucinactant 90 mg/kg — Administered via slow intra-tracheal instillation at a dose of 90 mg/kg (3.0 mL/kg of a 30-mg/mL suspension). Initial treatment given no later than 1 hour after randomization. Additional treatments were administered every 48 hours up to a maximum of 5 doses (up to DOL 18).
  Other Names: SURFAXIN; Lucinactant; Surfactant
  Arms: SURFAXIN Low Dose
Drug: Placebo — Sham air was administered via slow intratracheal instillation at a dose of 3.0 mL/kg volume of air. The initial treatment was given no later than 1 hour after randomization. Additional treatment were administered every 48 hours up to a maximum of 5 doses (up to DOL 18).
  Other Names: Sham Air
  Arms: Placebo

SUMMARY:
SURFAXIN® (lucinactant) treatment will be examined in very low birth weight infants to prevent development of chronic lung disease, commonly known as bronchopulmonary dysplasia (BPD), in premature infants who have required continued intubation and received surfactants for the prevention or treatment of respiratory distress syndrome (RDS).

DETAILED DESCRIPTION:
Determine the safety and tolerability of SURFAXIN administration in the first weeks of life as a therapeutic approach for prevention of BPD. Determine whether treatment with SURFAXIN during the first two to three weeks of life can decrease the proportion of infants on mechanical ventilation or oxygen or the incidence of death or BPD in VLBW infants when assessed at 28 days of life and 36 weeks post-menstrual age (as determined by the need for supplemental oxygen).

ELIGIBILITY:
Inclusion Criteria:

* Premature infants between 600 and 900 grams birth weight
* Intubated and on mechanical ventilation
* Sustained (>= 30 minutes) fraction of inspired oxygen (FiO₂) >= 0.30 within 8 hours prior to randomization

Exclusion Criteria:

* Mother has prolonged rupture of membranes ≥ 2 weeks
* Culture-proven sepsis
* High grade intraventricular hemorrhage (IVH)
* Congenital heart disease
* Congential anomalies inconsistent with life or likely to confound efficacy or safety endpoints
* FiO₂≥ 0.80 and mean airway pressure (MAP) ≥ 12 cmH2O at day of life (DOL) 3
* FiO₂< 0.25 at any time between meeting the entry criteria to immediately prior to randomization
* Concomitant use of any other surfactant within the first 48 hours of life
* Prior use of nitric oxide
* Prior use of steroids
* Current participation in any other clinical trial or has received an experimental drug or used an experimental device

Ages: 3 Days to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2005-02; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Guardia, MD, Study Director — Windtree Therapeutics; Matthew M Laughon, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Discovery Laboratories, Inc., Warrington, Pennsylvania, United States

REFERENCES:
- [Result] Laughon M, Bose C, Moya F, Aschner J, Donn SM, Morabito C, Cummings JJ, Segal R, Guardia C, Liu G; Surfaxin Study Group. A pilot randomized, controlled trial of later treatment with a peptide-containing, synthetic surfactant for the prevention of bronchopulmonary dysplasia. Pediatrics. 2009 Jan;123(1):89-96. doi: 10.1542/peds.2007-2680. PMID 19117865

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SURFAXIN High Dose | SURFAXIN Low Dose | Placebo
Started | 45 | 47 | 44
Completed | 44 | 47 | 44
Not Completed | 1 | 0 | 0
Not completed — Withdrew from study medication | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SURFAXIN High Dose | SURFAXIN Low Dose | Placebo | Total
Number analyzed (Participants) | 45 | 47 | 44 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 45 | 47 | 44 | 136
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 27 | 65
  Male | 24 | 30 | 17 | 71
Region of Enrollment [Number; unit: participants]
  United States | 17 | 20 | 19 | 56
  Chile | 8 | 10 | 7 | 25
  Poland | 17 | 14 | 16 | 47
  Hungary | 3 | 3 | 2 | 8
Gestational Age [Mean (Standard Deviation); unit: weeks] | 26.1 (1.68) | 25.5 (1.43) | 25.7 (1.36) | 25.8 (1.49)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Death or Bronchopulmonary Dysplasia (BPD) at 36 Weeks
Description: Number of participants who died or developed BPD, defined as oxygen requirement at 36 Weeks post-menstrual age
Time Frame: 36 weeks post-menstrual age (PMA)
Population: A sample size of 70 per arm is sufficient to demonstrate a 20% relative risk reduction. All randomized infants were analyzed (intent-to-treat)
Measure: Number; unit: participants
Arm/Group | SURFAXIN High Dose | SURFAXIN Low Dose | Placebo
Number analyzed (Participants) | 45 | 47 | 44
participants | 26 | 37 | 29
Statistical Analysis 1: Comparison: SURFAXIN High Dose vs Placebo; Null hypothesis: No difference between treatment groups; Test type: Superiority or Other; p = 0.476, Cochran-Mantel-Haenszel; Adjusting for pooled study center
Statistical Analysis 2: Comparison: SURFAXIN Low Dose vs Placebo; Null hypothesis: No difference between treatment groups; Test type: Superiority or Other; p = 0.208, Cochran-Mantel-Haenszel; Adjusting for pooled study center

2. Primary Outcome: All-cause Mortality
Time Frame: 36 weeks PMA
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SURFAXIN High Dose | SURFAXIN Low Dose | Placebo
Number analyzed (Participants) | 45 | 47 | 44
participants | 5 | 14 | 7
Statistical Analysis 1: Comparison: SURFAXIN High Dose vs Placebo; Null hypothesis: No difference between treatment groups; Test type: Superiority or Other; p = 0.500, Cochran-Mantel-Haenszel; Adjusting for pooled study center
Statistical Analysis 2: Comparison: SURFAXIN Low Dose vs Placebo; Null hypothesis: No difference between treatment groups; Test type: Superiority or Other; p = 0.146, Cochran-Mantel-Haenszel; Adjusting for pooled study center

3. Secondary Outcome: BPD at 28 Days
Description: BPD at 28 days of life, as determined by the need for supplemental oxygen
Time Frame: 28 days of life
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SURFAXIN High Dose | SURFAXIN Low Dose | Placebo
Number analyzed (Participants) | 45 | 47 | 44
participants | 42 | 44 | 38
Statistical Analysis 1: Comparison: SURFAXIN High Dose vs Placebo; Test type: Superiority or Other; p = 0.267, Cochran-Mantel-Haenszel; Adjusting for pooled study center
Statistical Analysis 2: Comparison: SURFAXIN Low Dose vs Placebo; Test type: Superiority or Other; p = 0.313, Cochran-Mantel-Haenszel; Adjusting for pooled study center
Statistical Analysis 3: Comparison: SURFAXIN High Dose vs SURFAXIN Low Dose; Test type: Superiority or Other; p = 0.944, Cochran-Mantel-Haenszel; Adjusting for pooled study center

4. Secondary Outcome: BPD at 36 Weeks
Description: BPD at 36 weeks PMA as determined by the need for supplemental oxygen
Time Frame: 36 weeks PMA
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SURFAXIN High Dose | SURFAXIN Low Dose | Placebo
Number analyzed (Participants) | 45 | 47 | 44
participants | 26 | 37 | 29
Statistical Analysis 1: Comparison: SURFAXIN High Dose vs Placebo; Test type: Superiority or Other; p = 0.476, Cochran-Mantel-Haenszel; Adjusting for pooled study center
Statistical Analysis 2: Comparison: SURFAXIN Low Dose vs Placebo; Test type: Superiority or Other; p = 0.208, Cochran-Mantel-Haenszel; Adjusting for pooled study center
Statistical Analysis 3: Comparison: SURFAXIN High Dose vs SURFAXIN Low Dose; Test type: Superiority or Other; p = 0.046, Cochran-Mantel-Haenszel; Adjusting for pooled study center

5. Secondary Outcome: Days Receiving Mechanical Ventilation (MV)
Description: Number of days receiving mechanical ventilation
Time Frame: 36 weeks PMA
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | SURFAXIN High Dose | SURFAXIN Low Dose | Placebo
Number analyzed (Participants) | 45 | 47 | 44
days | 30.1 (23.3) | 42.1 (26.4) | 35.8 (23.2)
Statistical Analysis 1: Comparison: SURFAXIN High Dose vs Placebo; Test type: Superiority or Other; p = 0.285, ANOVA; On rank adjusting for pooled study center
Statistical Analysis 2: Comparison: SURFAXIN Low Dose vs Placebo; Test type: Superiority or Other; p = 0.229, ANOVA; On rank adjusting for pooled study center
Statistical Analysis 3: Comparison: SURFAXIN High Dose vs SURFAXIN Low Dose; Test type: Superiority or Other; p = 0.030, ANOVA; On rank adjusting for pooled study center

6. Secondary Outcome: Duration of Supplemental Oxygen
Description: Number of days receiving supplemental oxygen through 36 weeks PMA
Time Frame: 36 weeks PMA
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | SURFAXIN High Dose | SURFAXIN Low Dose | Placebo
Number analyzed (Participants) | 45 | 47 | 44
days | 55.3 (16.8) | 63.0 (19.3) | 55.7 (23.4)
Statistical Analysis 1: Comparison: SURFAXIN High Dose vs Placebo; Test type: Superiority or Other; p = 0.483, ANOVA; On rank adjusting for pooled study center
Statistical Analysis 2: Comparison: SURFAXIN Low Dose vs Placebo; Test type: Superiority or Other; p = 0.123, ANOVA; On rank adjusting for pooled study center
Statistical Analysis 3: Comparison: SURFAXIN Low Dose; Test type: Superiority or Other; p = 0.006, ANOVA; On rank adjusting for pooled study center

7. Secondary Outcome: Area Under the Curve for Fraction of Inspired Oxygen (FiO₂)
Description: AUC for FiO₂calculated using the trapezoidal rule. Missing data imputed using last observation carried forward
Time Frame: 15 minutes prior to dose 1, 2 hours post dose 1, 6 hours post dose 1, 24 hours post dose 1, and daily from Study Day 2 to Study Day 25 and Day of Life 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent O₂*hour
Arm/Group | SURFAXIN High Dose | SURFAXIN Low Dose | Placebo
Number analyzed (Participants) | 45 | 47 | 44
Percent O₂*hour | 0.39 (0.14) | 0.41 (0.16) | 0.38 (0.17)
Statistical Analysis 1: Comparison: SURFAXIN High Dose vs Placebo; Test type: Superiority or Other; p = 0.843, ANOVA; Adjusting for pooled study center
Statistical Analysis 2: Comparison: SURFAXIN Low Dose vs Placebo; Test type: Superiority or Other; p = 0.543, ANOVA; Adjusting for pooled study center
Statistical Analysis 3: Comparison: SURFAXIN High Dose vs SURFAXIN Low Dose; Test type: Superiority or Other; p = 0.537, ANOVA; Adjusting for pooled study center

8. Secondary Outcome: Area Under the Curve for Mean Arterial Pressure (MAP)
Description: AUC for MAP (in mm Hg) calculated using the trapezoidal rule. Missing data imputed using last observation carried forward
Time Frame: 15 minutes prior to dose 1, 2 hours post dose 1, 6 hours post dose 1, 24 hours post dose 1, and daily from Study Day 2 to Study Day 25, and day of life 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: arterial pressure (mm Hg)*hour
Arm/Group | SURFAXIN High Dose | SURFAXIN Low Dose | Placebo
Number analyzed (Participants) | 45 | 47 | 44
arterial pressure (mm Hg)*hour | 5.99 (3.38) | 6.93 (4.13) | 6.34 (3.56)
Statistical Analysis 1: Comparison: SURFAXIN High Dose vs Placebo; Test type: Superiority or Other; p = 0.813, ANOVA; Adjusting for pooled study center
Statistical Analysis 2: Comparison: SURFAXIN Low Dose vs Placebo; Test type: Superiority or Other; p = 0.449, ANOVA; Adjusting for pooled study center
Statistical Analysis 3: Comparison: SURFAXIN High Dose vs SURFAXIN Low Dose; Test type: Superiority or Other; p = 0.275, ANOVA; Adjusting for pooled study center

9. Secondary Outcome: Incidence of Death or BPD at 28 Days
Description: Death or BPD, defined as oxygen requirement at 28 days of life
Time Frame: 28 days of life
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SURFAXIN High Dose | SURFAXIN Low Dose | Placebo
Number analyzed (Participants) | 45 | 47 | 44
participants | 42 | 44 | 38
Statistical Analysis 1: Comparison: SURFAXIN High Dose vs Placebo; Test type: Superiority or Other; p = 0.267, Cochran-Mantel-Haenszel; Adjusting for pooled study center
Statistical Analysis 2: Comparison: SURFAXIN Low Dose vs Placebo; Test type: Superiority or Other; p = 0.313, Cochran-Mantel-Haenszel; Adjusting for pooled study center

10. Secondary Outcome: Days in Hospital
Description: The number of days spent in the hospital through 36 weeks PMA
Time Frame: 36 weeks PMA
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | SURFAXIN High Dose | SURFAXIN Low Dose | Placebo
Number analyzed (Participants) | 45 | 47 | 44
days | 65.8 (11.72) | 70.0 (10.06) | 68.6 (9.57)
Statistical Analysis 1: Comparison: SURFAXIN High Dose vs Placebo; Test type: Superiority or Other; p = 0.311, ANOVA; On rank adjusting for pooled study center
Statistical Analysis 2: Comparison: SURFAXIN Low Dose vs Placebo; Test type: Superiority or Other; p = 0.516, ANOVA; On rank adjusting for pooled study center
Statistical Analysis 3: Comparison: SURFAXIN High Dose vs SURFAXIN Low Dose; Test type: Superiority or Other; p = 0.094, ANOVA; On rank adjusting for pooled study center

ADVERSE EVENTS:
Time Frame: Through 36 weeks PMA
Arm/Group | SURFAXIN High Dose | SURFAXIN Low Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 33/45 | 36/47 | 35/44
Other Adverse Events (participants affected / at risk) | 45/45 | 47/47 | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SURFAXIN High Dose (N=45) | SURFAXIN Low Dose (N=47) | Placebo (N=44)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia NOS (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2)
Cardiac arrest neonatal (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest neonatal (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 3 (3) | 3 (3) | 1 (1)
Retrolental fibro-dysplasia (Eye disorders) | 8 (8) | 9 (9) | 8 (8)
Ileal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Inguinal hernia NOS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal perforation NOS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Meconium ileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Necrotising enterocolitis (Gastrointestinal disorders) | 4 (4) | 5 (5) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchopneumonia NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neonatal meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia NOS (Infections and infestations) | 1 (1) | 1 (1) | 1 (2)
Sepsis NOS (Infections and infestations) | 4 (4) | 0 (0) | 1 (1)
Sepsis neonatal (Infections and infestations) | 3 (3) | 6 (6) | 6 (6)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septicaemia serratia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septicaemia staphylococcal (Infections and infestations) | 4 (4) | 5 (5) | 4 (4)
Abrasion NOS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 2 (2) | 4 (8) | 2 (2)
Diabetes mellitus NOS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis NOS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Convulsions NOS (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Hydrocephalus NOS (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 3 (3) | 3 (3) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure neonatal (Renal and urinary disorders) | 0 (0) | 5 (5) | 1 (1)
Urinary tract infection NOS neonatal (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Atelectasis neonatal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (8) | 9 (9)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 0 (0)
Neonatal apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2)
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 1 (1) | 0 (0)
Neonatal respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 5 (5) | 3 (3)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
Pulmonary interstitial emphysema syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Patent ductus arteriosus repair (Surgical and medical procedures) | 7 (7) | 8 (8) | 8 (8)
Circulatory failure neonatal (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Intracranial haemorrhage NOS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Intraventricular haemorrhage neonatal (Vascular disorders) | 4 (4) | 9 (9) | 7 (8)
Neonatal hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SURFAXIN High Dose (N=45) | SURFAXIN Low Dose (N=47) | Placebo (N=44)
Anaemia NOS (Blood and lymphatic system disorders) | 10 (27) | 6 (8) | 8 (20)
Anaemia neonatal (Blood and lymphatic system disorders) | 24 (41) | 25 (37) | 25 (38)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 5 (5)
Thrombocytopenia neonatal (Blood and lymphatic system disorders) | 6 (6) | 7 (8) | 10 (10)
Bradycardia NOS (Cardiac disorders) | 16 (29) | 20 (51) | 8 (11)
Neonatal tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 3 (3)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 14 (15) | 11 (13) | 16 (16)
Hypothyroidism (Endocrine disorders) | 3 (3) | 2 (2) | 4 (4)
Retrolental fibro-dysplasia (Eye disorders) | 27 (30) | 29 (35) | 29 (35)
Gastro-oesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 12 (12) | 9 (9)
Inguinal hernia NOS (Gastrointestinal disorders) | 5 (7) | 7 (7) | 4 (4)
Necrotising enterocolitis (Gastrointestinal disorders) | 8 (8) | 10 (10) | 5 (5)
Oedema NOS (General disorders) | 2 (2) | 1 (1) | 7 (7)
Cholestasis (Hepatobiliary disorders) | 3 (3) | 2 (2) | 6 (6)
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 (4) | 3 (3) | 8 (8)
Hypoproteinaemia (Hepatobiliary disorders) | 2 (2) | 2 (2) | 4 (4)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2) | 3 (4)
Pneumonia NOS (Infections and infestations) | 7 (7) | 6 (6) | 4 (6)
Sepsis NOS (Infections and infestations) | 4 (5) | 3 (3) | 3 (5)
Sepsis Neonatal (Infections and infestations) | 7 (8) | 17 (19) | 12 (15)
Septicaemia staphylococcal (Infections and infestations) | 13 (14) | 13 (14) | 14 (15)
Tracheitis NOS (Infections and infestations) | 2 (2) | 5 (8) | 3 (5)
Urinary tract infection fungal (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Abrasion NOS (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 6 (6)
Blood in stool (Investigations) | 3 (3) | 1 (1) | 3 (3)
Oxygen saturation decreased (Investigations) | 17 (42) | 18 (40) | 16 (22)
Acidosis NOS (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 3 (3)
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 10 (11) | 9 (11) | 7 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (4)
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (5) | 3 (3) | 5 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (14) | 15 (19) | 13 (15)
Metabolic acidosis NOS (Metabolism and nutrition disorders) | 4 (4) | 9 (11) | 9 (9)
Osteopenia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 3 (3)
Convulsions NOS (Nervous system disorders) | 4 (4) | 6 (6) | 8 (10)
Neurological disorder NOS (Nervous system disorders) | 5 (5) | 3 (3) | 2 (2)
Renal failure neonatal (Renal and urinary disorders) | 2 (2) | 8 (8) | 6 (6)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (7) | 3 (3)
Atelectasis neonatal (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 3 (3)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 39 (39) | 34 (36) | 37 (38)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 6 (9) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (13) | 4 (5) | 2 (2)
Neonatal apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 18 (20) | 14 (16)
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 18 (41) | 25 (75) | 7 (10)
Neonatal respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 5 (5) | 2 (2)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 1 (1) | 2 (2)
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 7 (7) | 3 (3)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 6 (6)
Pulmonary interstitial emphysema syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 7 (7)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (2) | 3 (3)
Respiratory failure (exc neonatal) (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 4 (4)
Patent ductus arteriosus repair (Surgical and medical procedures) | 8 (8) | 8 (8) | 8 (8)
Hypertension neonatal (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Intraventricular haemorrhage neonatal (Vascular disorders) | 17 (18) | 25 (26) | 17 (19)
Neonatal hypotension (Vascular disorders) | 5 (5) | 8 (8) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes